CLINICAL TRIAL: NCT05488392
Title: Safety and Tolerability of Intrajugular Cooling in Patients With Acute Ischemic Stroke After Mechanical Thrombectomy
Brief Title: Hypothermia With Intrajugular Cooling in Acute Ischemic Stroke Thrombectomy
Acronym: PICNIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PICNIC
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; hypothermia; thrombectomy; intrajugular cooling
MeSH Terms: conditions — Ischemic Stroke; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrajugular cooling group (Experimental): The safety and tolerability of hypothermia with intrajugular cooling will be investigated using 3+3 dose-escalation trial design.
  Interventions: Procedure: Hypothermia with intrajugular cooling

INTERVENTIONS:
Procedure: Hypothermia with intrajugular cooling — Hypothermia with intrajugular cooling will be applied after successful recanalization of the culprit internal carotid artery/middle cerebral artery. The perfusion rate will be set at 30 ml/min. Low temperature saline will be infused into the internal jugular vein for 10 min, 15 min, 20 min, 25 min, and 30 min successively.

SUMMARY:
Hypothermia with intrajugular cooling is a neuroprotective strategy that has been proven to minimize brain damage and maximize functional preservation in animal models of stroke. The purpose of this proof-of-concept study is to determine the safety and tolerability of intrajugular cooling in patients with acute ischemic stroke who are treated with mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. Acute ischemic stroke caused by unilateral internal carotid artery terminal segment/middle cerebral artery M1 segment occlusion;
3. In line with the indications for mechanical thrombectomy without contraindications;
4. Successful recanalization (mTICI 2b/3) after mechanical thrombectomy that confirmed by digital subtraction angiography;
5. Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

1. Suffering from cerebral venous system diseases such as cerebral venous thrombosis/stenosis/dysplasia;
2. Suffering from heart diseases such as ventricular arrhythmia/myocardial infarction/congestive heart failure;
3. Imaging examination after mechanical thrombectomy shows intracranial hemorrhage/contrast extravasation;
4. Difficulty in reaching the designated position of the device used for intrajugular cooling;
5. Difficulty in complying with intrajugular cooling or other conditions that the investigator considered inappropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major response | Within 24 hours after hypothermia with intrajugular cooling
  Major response is any of the following:
  1. Cerebral venous system damage;
  2. Cerebral venous thrombosis;
  3. Huge hematoma at the puncture site requiring surgical intervention;
  4. Malignant arrhythmia within 24 hours;
  5. Cardiac arrest within 24 hours;
  6. Myocardial infarction within 24 hours;
  7. Congestive heart failure within 24 hours.
  In the 3 + 3 design, 3 subjects are recruited for a given intrajugular cooling dose level. The trial is stopped if ≥ 2 of 3 subjects at a given dose level show major response. If only 1 of 3 subjects shows major response, 3 more subjects are recruited at a given dose level and a major response in any of them will stop the trial. Otherwise, same procedure is followed for the next dose level. Maximum tolerable dose will be the dose at the level before stopping of the trial. The schedule of advancing duration is 10 min, 15 min, 20 min, 25 min, and 30 min.

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.